CLINICAL TRIAL: NCT04628260
Title: UNCOVER - a Non-interventional Study to Investigate Undiagnosed Severe Asthma
Status: Completed | Type: Observational
Sponsor: Karl Landsteiner Institute for Clinical and Experimental Pneumology (Other)
Collaborators: Universitätsklinik für Innere Medizin II, Pulmologie (Unknown)
Responsible Party: Sponsor
Other Study IDs: 213799
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
UNCOVER is a non-interventional study to investigate the prevalence of difficult-to-treat and severe Asthma eligible for treatment with biologics in a cohort of patients with suspected, so far undiagnosed severe Asthma which were previously treated by General practitioners and Office-based pulmonologists.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at inclusion
* written informed consent
* currently diagnosed with Asthma fulfilling at least one of the criteria of potential severe Asthma
* willing and able to complete the study questionnaire miniAQLQ

Exclusion Criteria:

* biological Treatment for Asthma during the past 12 months
* participation in a clinical Trial within the last 3 months
* patients who are not able to read or write, who do not understand the nature of the study or the ICF or who are dependent from the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male patients are eligible for this non-interventional study when fulfilling all criteria for inclusion and None of the criteria for exclusion. 400 patients will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The Primary objective is the Investigation of the prevalence of difficult-to-treat and severe Asthma eligible for Treatment with biologics. | 18 months
  Number of patients with diagnosis of severe Asthma according to the ATS/ERS Definition of severe Asthma and number of severe Asthma patients eligible for one or more biologic Treatments for Asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Pohl, Univ. Prof. Dr., Principal Investigator — Head of Karl Landsteiner Institut for Clinical and Experimental Pneumology
Locations (1):
- Karl Landsteiner Institute for Clinical and Experimental Pneumology, Klinik Hietzing, Vienna, Austria